CLINICAL TRIAL: NCT06293508
Title: mHealth Behavioural Intervention to Increase Breast Cancer Screening Rates Among Members of the Public
Acronym: mBLISS-B
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Project was halted due to administrative complications arising while seeking for a vendor to assist with subject recruitment.
Sponsor: Clinical Research Centre, Malaysia (Other)
Collaborators: Ministry of Health, Malaysia (Other Government); National University of Malaysia (Other); Institute for Health Behavioral Research, Malaysia (Unknown)
Responsible Party: Principal Investigator, Nicholas Hing Yee Liang, Principal Investigator, Clinical Research Centre, Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: NMRR ID-22-02616-I2I
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Breast Neoplasm Female
Keywords: mHealth; breast cancer screening; behaviour; health communication; randomised controlled trial; behaviour change communication; persuasive communication; social messaging
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (No Intervention): Participants do not receive any message throughout the study period.
- Experimental Arm 1 (Experimental): Participants in this group will receive a message on a weekly basis throughout the intervention period, which is 6 months, via WhatsApp.
  Interventions: Behavioral: Standard Health Communication Intervention
- Experimental Arm 2 (Experimental): Participants in this group will receive a message on a weekly basis throughout the intervention period, which is 6 months, via WhatsApp.
  Interventions: Behavioral: Behavioural Change Health Communication Intervention

INTERVENTIONS:
Behavioral: Standard Health Communication Intervention — Participants in this group will receive links and materials related to breast cancer screening from official sources (e.g. MOH, Non-governmental organizations (NGOs), etc.) that is already readily available and accessible by the Malaysian public. Frequency, duration, and platform of dissemination will be based on findings from Phase 1 of this study.
  Arms: Experimental Arm 1
Behavioral: Behavioural Change Health Communication Intervention — Participants receive health communication materials designed using persuasive behavioural change communication principles and behavior science to promote breast cancer screening. Frequency, duration, and platform of dissemination will be based on findings from Phase 1 of this study.
  Arms: Experimental Arm 2

SUMMARY:
Late-stage presentation of breast cancer cases are on the rise in Malaysia. Encouraging breast screening practices can assist in early breast cancer detection. Literature has proven that behavior interventions in the form of behavior change health communication using social messaging applications is a viable strategy and potentially effective at motivating breast cancer screening among the public. Such studies are scarce in the South East Asian region, particularly in Malaysia, which is the prime motivation for the current study,

Based on this promising prospect, a randomized controlled trial will be designed to study the effects of applying persuasive health communication materials to initiate behavior change among a group of Malaysian women. Materials are delivered in the form of a health communication program over a social messaging application to promote breast cancer screening practices, which is either a clinical breast examination, or a mammogram. The investigators hypothesize that Malaysian women who are exposed to such materials that are designed based on behavior science and behavior change principles will be nudged and hence more likely to attend breast cancer screening compared to a control group.

DETAILED DESCRIPTION:
This study involves a randomized controlled trial to asses the effectiveness of a health communication program using specifically designed materials using behavior science and behavior change principles. Materials were designed based on findings derived from a scoping review and interviewing Malaysian women through a series of qualitative interviews to determine the barriers and facilitators of attending breast cancer screening. The interview also investigated women's preferences for certain characteristics in a health message and health communication program that would motivate them to attend screening.

Participants in the main experimental group will be compared with a control group, and another group which undergoes a standard health communication program.

ELIGIBILITY:
Inclusion Criteria:

1. Malaysian women aged 40 years and above
2. Possess a smartphone with the predetermined social messaging application (derived from Phase 1 of study) installed.
3. Have not been diagnosed with cancer before.

Exclusion Criteria:

1. Underwent Clinical Breast Examination in the past 12 months.
2. Mammogram screening in the past 2 years.
3. Subjects who are deemed to have cognitive impairment and unable to provide consent to the study.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1180 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Breast cancer screening attendance (either clinical breast examination (CBE) or mammogram). | 2 time points: 3 months after 6 month intervention period has ended, and 6 months after 6 month intervention period has ended.
  Self-reported attendance of breast cancer screening

SECONDARY OUTCOMES:
Health literacy level | At baseline
  Scored via a validated instrument
Perception based on domains in Health Belief Model | 3 time points: Baseline, 3 months after 6 month intervention period has ended, and 6 months after 6 month intervention period has ended.
  Scored via a validated revised Champion Health Belief Model Scale instrument
Perceived acceptance and usefulness of health communication program | 3 months after 6 month intervention period has ended.
  Scored via a validated instrument
Reasons behind participants not participating in breast cancer screening. | 2 time points: Baseline, and 3 months after 6 month intervention period has ended.
  Determined via a multiple choice question

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Yee Liang Hing, MSc, Principal Investigator — Institute for Clinical Research, National Institutes of Health, Malaysia
Locations (1):
- Institute for Clinical Research, National Institutes of Health, Malaysia, Shah Alam, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD.